CLINICAL TRIAL: NCT04010344
Title: Addressing Hypertension Control in Africa (ADHINCRA) Study
Brief Title: Addressing Hypertension Care in Africa
Acronym: ADHINCRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Johns Hopkins Alliance for a Healthier World (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00218586
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Hypertension; Diabetes; Telemedicine
MeSH Terms: conditions — Hypertension; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Two-arm pilot cluster randomized control trial involving 240 participants with uncontrolled hypertension. The healthcare setting is the unit of randomization and patients are the unit of analysis. Each of the four healthcare settings will be recruited and randomly assigned to the multilevel intervention or control group. Randomization will be performed using a computer-generated random sequence program with a 1:1 allocation and a block size of 6 (to assure equal numbers in each arm). After meeting the study criteria for enrollment, 60 eligible patients for each setting will be assigned to either control or intervention arm according to their healthcare setting's intervention assignment by the study coordinator. The intervention will be administered for six months following which it will be withdrawn, and patients will be followed for six more months to assess outcomes.
Who Masked: Participant, Outcomes Assessor
Masking Description: Other staff will conduct the evaluations using established protocols. They will remain blinded as to patients' group status throughout the study (i.e., pre-intervention, 1, 3, 6 & 9-month evaluations).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care Group (Experimental): All participants in the enhanced usual care arm must own a cell phone with at least short message service (SMS) and voicemail. To control for attention exposure, they will receive SMS messages daily dealing with healthy lifestyle behaviors (smoking, diet, physical activity) but not with medication adherence or hypertension-specific issues. Every three days (comparable to intervention group monitoring) they will receive an automated SMS directing them to a different 2-3 min video/YouTube™ clips on healthy lifestyles. Patients in this arm of the study will also receive usual care as determined by their providers. Usual care is described in the next section.
  Interventions: Behavioral: Enhanced Usual Care Group
- Usual Care (Active Comparator): Patients in this arm of the study will receive usual care as determined by their providers. Usual care in the region typically involves at least one visit every 2-3 months for review of adherence to treatment, blood pressure control, and prescriptions for medication refills. Similar to the intervention group, participants will have a total of three follow-up visits which will be separate from their regular appointments during which study outcomes will be assessed.
  Interventions: Other: Usual Care Group

INTERVENTIONS:
Behavioral: Enhanced Usual Care Group — Medtronic® Labs' Akoma pa app, a culturally-tested and locally attuned mobile health platform, will be used in the intervention arm of the study to improve communication between the Community Health Officer (CHO) and the participant. This platform will be used to enhance shared decision making, clinical decision support, participatory communication, knowledge, treatment adherence (medication and lifestyle modification), and self-monitoring of hypertension. We will test the feasibility of the Akoma pa app in addressing patient-level and provider-level barriers to hypertension control.
  The app will consist of the following components:
  1. Reminders
  2. Participant to CHO messaging
  3. Home BP tracking
  4. Educational materials on cardiovascular disease (CVD) and Stroke- Participants will have access to education modules on reducing the risk of CVD and stroke tailored to their knowledge level.
  5. CHO provider portal- The provider portal will include decision support tools.
  Arms: Enhanced Usual Care Group
Other: Usual Care Group — Regular/usual appointments or visits to patients' healthcare provider for management of study outcomes
  Arms: Usual Care

SUMMARY:
A pilot cluster randomized control trial to test the feasibility of a multilevel, nurse-led, mobile health enhanced intervention in patients with uncontrolled hypertension in Ghana

DETAILED DESCRIPTION:
This is a two-arm pilot cluster randomized controlled trial (RCT) involving 240 participants with uncontrolled hypertension (HTN) with the healthcare setting as the unit of randomization and patients as the unit of analysis. Each of the four healthcare settings will be recruited and randomly assigned to the multilevel intervention or control group. A statistician will generate the randomization using a computer-generated random sequence program with an allocation ratio of 1:1 and a block size of 6 (to assure equal numbers in each arm). After having met study criteria for enrollment, 60 eligible patients for each setting will be assigned to either control or intervention arm according to the patients' healthcare setting's intervention assignment by the study coordinator. A cluster RCT has been chosen to avoid potential treatment contamination in which physicians within healthcare settings might unintentionally provide patients with different degrees of attention or blending of treatment protocols. The intervention will be administered for six months following which it will be withdrawn, and patients will be followed for six more months to assess outcomes.

The investigators will use quota sampling to over sample socioeconomically deprived persons to ensure that socioeconomically deprived persons comprise 50% of the sample. Poverty will be defined by (1) Household income, based on Ghana minimum monthly wage of 210 Ghana cedis (equivalent of $55). After screening eligible participants, the investigators will assign four clusters of 60 patients to the intervention or control arms. The investigators will require 30 patients in each cluster to be male and 30 to be female since in the investigators' previous work, men have been underrepresented potentially due to gender-differences in healthcare seeking behaviors. Men have also had inferior treatment and control rates in previous studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if they are 18-70 years old;
* Male or female
* Uncontrolled hypertension (SBP ≥140 mm Hg) based upon last outpatient encounter within the previous three months
* Patients with previous strokes, coronary artery disease, up to stage three kidney disease and diabetes mellitus meeting BP cut-off criteria will be eligible for enrollment.

Exclusion Criteria:

* Patients will be excluded if they fail to meet any of the above inclusion criteria
* Severe cognitive impairment/dementia (Modified Mini-Mental State Examination (MMSE) score ≤24)
* Severe global disability (modified Rankin Scale (mRS) score ≥3)
* Not able to independently follow blood pressure measurement protocol or use of Smartphone for study protocol or without a care-giver to assist with BP monitoring at home
* Patients with estimated glomerular filtration rate (eGFR) <30ml/min

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2019-07-14 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Blood Pressure levels from Baseline | Baseline, 1 month , 3 months, 6 months, 9 months, 12 months
  Changes in Blood pressure levels, measured in mmHg, will be assessed at the baseline, 1-month, 3-month, 6-month, 9-month, and 12-month visits.
Change in Blood Pressure control by poverty status from Baseline | Baseline, 1 month , 3 months, 6 months, 9 months, 12 months
  Blood pressure control - defined as systolic blood pressure (SBP) < 140 mm Hg SBP reduction will be compared by deprivation status defined by monthly income < 210 Ghana cedis determined at the enrollment visit.

SECONDARY OUTCOMES:
Change in glycohemoglobin (A1C) between arms | Baseline, 1 month , 3 months, 6 months, 9 months, 12 months
  Hgb A1C in both study arms will be examined for change at the 1-month, 3-month, 6-month, 9-month, and 12-month visits after the initial baseline assessment.
Difference in Hypertensive Urgencies and Emergencies between arms | Baseline, 1 month , 3 months, 6 months, 9 months, 12 months
  Difference in the number of emergency room visits (for hypertensive urgencies and/or emergencies) for both arms will be examined at the 1-month, 3-month, 6-month, 9-month, and 12-month visits. after the initial baseline assessment.
Difference in Cardiovascular Disease (CVD) Events between study arms | Baseline, 1 month , 3 months, 6 months, 9 months, 12 months
  Difference in the number of CVD events (such as strokes, coronary artery disease, heart failures, and deaths) for both arms will be examined at the 1-month, 3-month, 6-month, 9-month, and 12-month visits after the initial baseline assessment.
Difference in treatment adherence as assessed by the Hill-Bone Medication Adherence Scale | At 6 months
  Self-Reported Medication Adherence will be assessed with the 9-item Hill-Bone Medication Adherence Scale and compared in both arms at months 6 and 12 by poverty status. The Hill-Bone has broad applicability in measuring medication adherence in patients with hypertension, diabetes, chronic obstructive pulmonary disease, stroke among others. Scores range from 9 - 36 with higher scores indicating poorer adherence to antihypertensive drug therapy.
Difference in treatment adherence as assessed by the Hill-Bone Medication Adherence Scale | At 12 months
  Self-Reported Medication Adherence will be assessed with the 9-item Hill-Bone Medication Adherence Scale and compared in both arms at months 6 and 12 by poverty status. The Hill-Bone has broad applicability in measuring medication adherence in patients with hypertension, diabetes, chronic obstructive pulmonary disease, stroke among others. Scores range from 9 - 36 with higher scores indicating poorer adherence to antihypertensive drug therapy.
Change in the acceptability and usability of the Akoma pa app score as assessed by the Marshfield System Usability Survey | At 1 month , 3 months, 6 months, 9 months, 12 months
  The acceptability and usability of the Akoma pa app will be assessed with the 16-item Marshfield System Usability Survey. Scores on this instrument range from 16 to 80 with higher scores indicating better usability. This will be examined at the 1-month, 3-month, 6-month, 9-month, and 12-month visits after the initial baseline assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Commodore-Mensah, PhD, MHS, RN, Principal Investigator — Johns Hopkins University
Locations (4):
- Ghana (4):
  - Komfo Anokye Teaching Hospital, Kumasi, Ashanti Region
  - Kumasi South Hospital, Kumasi, Ashanti Region
  - Manhyia Government Hospital, Kumasi, Ashanti Region
  - Suntreso Government Hospital, Kumasi, Ashanti Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kearney PM, Whelton M, Reynolds K, Muntner P, Whelton PK, He J. Global burden of hypertension: analysis of worldwide data. Lancet. 2005 Jan 15-21;365(9455):217-23. doi: 10.1016/S0140-6736(05)17741-1. PMID 15652604
- [Background] Sarfo-Kantanka O, Sarfo FS, Oparebea Ansah E, Eghan B, Ayisi-Boateng NK, Acheamfour-Akowuah E. Secular Trends in Admissions and Mortality Rates from Diabetes Mellitus in the Central Belt of Ghana: A 31-Year Review. PLoS One. 2016 Nov 22;11(11):e0165905. doi: 10.1371/journal.pone.0165905. eCollection 2016. PMID 27875539
- [Background] Sarfo FS, Ovbiagele B, Gebregziabher M, Wahab K, Akinyemi R, Akpalu A, Akpa O, Obiako R, Owolabi L, Jenkins C, Owolabi M; SIREN. Stroke Among Young West Africans: Evidence From the SIREN (Stroke Investigative Research and Educational Network) Large Multisite Case-Control Study. Stroke. 2018 May;49(5):1116-1122. doi: 10.1161/STROKEAHA.118.020783. Epub 2018 Apr 4. PMID 29618553
- [Background] Staessen JA, Wang JG, Thijs L. Cardiovascular protection and blood pressure reduction: a meta-analysis. Lancet. 2001 Oct 20;358(9290):1305-15. doi: 10.1016/S0140-6736(01)06411-X. PMID 11684211
- [Background] Agyemang C, Nyaaba G, Beune E, Meeks K, Owusu-Dabo E, Addo J, Aikins AD, Mockenhaupt FP, Bahendeka S, Danquah I, Schulze MB, Galbete C, Spranger J, Agyei-Baffour P, Henneman P, Klipstein-Grobusch K, Adeyemo A, van Straalen J, Commodore-Mensah Y, Appiah LT, Smeeth L, Stronks K. Variations in hypertension awareness, treatment, and control among Ghanaian migrants living in Amsterdam, Berlin, London, and nonmigrant Ghanaians living in rural and urban Ghana - the RODAM study. J Hypertens. 2018 Jan;36(1):169-177. doi: 10.1097/HJH.0000000000001520. PMID 28858173
- [Background] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Background] Sanuade OA, Awuah RB, Kushitor M. Hypertension awareness, treatment and control in Ghana: a cross-sectional study. Ethn Health. 2020 Jul;25(5):702-716. doi: 10.1080/13557858.2018.1439898. Epub 2018 Feb 15. PMID 29448808
- [Background] Sarfo FS, Mobula LM, Burnham G, Ansong D, Plange-Rhule J, Sarfo-Kantanka O, Ofori-Adjei D. Factors associated with uncontrolled blood pressure among Ghanaians: Evidence from a multicenter hospital-based study. PLoS One. 2018 Mar 19;13(3):e0193494. doi: 10.1371/journal.pone.0193494. eCollection 2018. PMID 29554106
- [Background] Commodore-Mensah Y, Samuel LJ, Dennison-Himmelfarb CR, Agyemang C. Hypertension and overweight/obesity in Ghanaians and Nigerians living in West Africa and industrialized countries: a systematic review. J Hypertens. 2014 Mar;32(3):464-72. doi: 10.1097/HJH.0000000000000061. PMID 24445390
- [Background] Stephenson J. Noncompliance may cause half of antihypertensive drug "failures". JAMA. 1999 Jul 28;282(4):313-4. doi: 10.1001/jama.282.4.313. No abstract available. PMID 10432015
- [Background] Kretchy IA, Owusu-Daaku FT, Danquah S. Locus of control and anti-hypertensive medication adherence in Ghana. Pan Afr Med J. 2014 Jan 18;17 Suppl 1(Suppl 1):13. doi: 10.11694/pamj.supp.2014.17.1.3433. eCollection 2014. PMID 24624246
- [Background] Ogedegbe G, Plange-Rhule J, Gyamfi J, Chaplin W, Ntim M, Apusiga K, Iwelunmor J, Awudzi KY, Quakyi KN, Mogaverro J, Khurshid K, Tayo B, Cooper R. Health insurance coverage with or without a nurse-led task shifting strategy for hypertension control: A pragmatic cluster randomized trial in Ghana. PLoS Med. 2018 May 1;15(5):e1002561. doi: 10.1371/journal.pmed.1002561. eCollection 2018 May. PMID 29715303
- [Background] Barry MJ, Edgman-Levitan S. Shared decision making--pinnacle of patient-centered care. N Engl J Med. 2012 Mar 1;366(9):780-1. doi: 10.1056/NEJMp1109283. No abstract available. PMID 22375967
- [Background] Bakken S, Grullon-Figueroa L, Izquierdo R, Lee NJ, Morin P, Palmas W, Teresi J, Weinstock RS, Shea S, Starren J; IDEATel Consortium. Development, validation, and use of English and Spanish versions of the telemedicine satisfaction and usefulness questionnaire. J Am Med Inform Assoc. 2006 Nov-Dec;13(6):660-7. doi: 10.1197/jamia.M2146. Epub 2006 Aug 23. PMID 16929036
- [Background] Demiris G, Speedie S, Finkelstein S. A questionnaire for the assessment of patients' impressions of the risks and benefits of home telecare. J Telemed Telecare. 2000;6(5):278-84. doi: 10.1258/1357633001935914. PMID 11070589
- [Background] Lakshminarayan K, Westberg S, Northuis C, Fuller CC, Ikramuddin F, Ezzeddine M, Scherber J, Speedie S. A mHealth-based care model for improving hypertension control in stroke survivors: Pilot RCT. Contemp Clin Trials. 2018 Jul;70:24-34. doi: 10.1016/j.cct.2018.05.005. Epub 2018 May 12. PMID 29763657
- [Background] Glasgow RE, McKay HG, Piette JD, Reynolds KD. The RE-AIM framework for evaluating interventions: what can it tell us about approaches to chronic illness management? Patient Educ Couns. 2001 Aug;44(2):119-27. doi: 10.1016/s0738-3991(00)00186-5. PMID 11479052
- [Derived] Commodore-Mensah Y, Sarfo FS, Turkson-Ocran RA, Foti K, Mobula LM, Himmelfarb CD, Carson KA, Appiah LT, Degani M, Lang'at C, Nyamekye G, Molello NE, Ahima R, Cooper LA. Addressing Hypertension Care in Africa (ADHINCRA): Study protocol for a cluster-randomized controlled pilot trial. Contemp Clin Trials. 2023 Feb;125:107077. doi: 10.1016/j.cct.2022.107077. Epub 2022 Dec 30. PMID 36592818
- See also: World Health Organization(WHO). Chapter XIII: Hypertension in adherence to LongTerm therapies-evidence for action. — http://apps.who.int/iris/bitstream/handle/10665/42682/9241545992.pdf?sequence=1
- See also: World Health Statistics — http://www.who.int/gho/publications/world_health_statistics/2015/en/